CLINICAL TRIAL: NCT07235007
Title: Survival Impact of Repeated Endobiliary Radiofrequency Ablation in Patients Undergoing Durvalumab Plus Gemcitabine and Cisplatin for Extrahepatic Cholangiocarcinoma: An International Multicenter Randomized Controlled Trial (BRAVE Trial)
Brief Title: Repeated Endobiliary Radiofrequency Ablation Plus Durvalumab, Gemcitabine, and Cisplatin for Unresectable Extrahepatic Cholangiocarcinoma
Acronym: BRAVE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aichi Medical University (Other)
Responsible Party: Principal Investigator, Tadahisa Inoue, Associate Professor, Aichi Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BRAVE-001
Record Dates: First submitted 2025-11-16; First posted 2025-11-19 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-11

CONDITIONS: Extrahepatic Cholangiocarcinoma
Keywords: Extrahepatic Cholangiocarcinoma; Cholangiocarcinoma; Biliary Tract Cancer; Bile Duct Stricture; Endobiliary Radiofrequency Ablation (EB-RFA); Radiofrequency Ablation; Endoscopic Retrograde Cholangiopancreatography (ERCP); Gemcitabine; Cisplatin; Durvalumab; Recurrent Biliary Obstruction (RBO)
MeSH Terms: conditions — Cholangiocarcinoma; Biliary Tract Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endobiliary Radiofrequency Ablation + Plastic Stent + Durvalumab/Gemcitabine/Cisplatin (Experimental): Participants undergo endobiliary radiofrequency ablation (EB-RFA) followed by placement of a plastic biliary stent during the index endoscopy. A scheduled second endoscopy at Month 3 (window 2-4 months) includes repeat EB-RFA and stent exchange. Additional EB-RFA sessions (≥2-month intervals) may be performed if imaging suggests a potentially ablatable residual biliary lesion. All participants receive systemic therapy with durvalumab, gemcitabine, and cisplatin according to institutional standards.
  Interventions: Device: Endobiliary Radiofrequency Ablation (EB-RFA); Device: Plastic Biliary Stent
- Plastic Stenting + Durvalumab/Gemcitabine/Cisplatin (Active Comparator): Participants receive standard endoscopic placement of a plastic biliary stent during the index endoscopy without EB-RFA. A scheduled elective stent exchange is performed at Month 3 (window 2-4 months). Additional elective stent exchanges every ≥2 months may be performed at the investigator's discretion. All participants receive systemic therapy with durvalumab, gemcitabine, and cisplatin according to institutional standards.
  Interventions: Device: Plastic Biliary Stent

INTERVENTIONS:
Device: Endobiliary Radiofrequency Ablation (EB-RFA) — Endobiliary RFA performed using the ELRA® catheter (STARmed) with VIVA combo® generator.
  Recommended settings: 7-10 W, temperature control 80 °C, 120 seconds per application.
  Applied along the full stricture length. Repeat procedure at Month 3 (window 2-4 months).
  Additional sessions every ≥2 months permitted if imaging suggests ablatable residual lesion.
  Arms: Endobiliary Radiofrequency Ablation + Plastic Stent + Durvalumab/Gemcitabine/Cisplatin
Device: Plastic Biliary Stent — Placement of 7Fr or 8.5Fr plastic biliary stent from hepatic side of the stenosis to the duodenum.
  Bilateral preferred for hilar strictures; unilateral acceptable based on drainage.

SUMMARY:
This international, multicenter, open-label randomized controlled trial evaluates whether repeated endobiliary radiofrequency ablation (EB-RFA) improves overall survival in patients with unresectable extrahepatic cholangiocarcinoma undergoing first-line systemic therapy with durvalumab plus gemcitabine and cisplatin (GCD). Eligible patients will be randomized 1:1 to EB-RFA with plastic stent placement or standard plastic stenting alone. A scheduled second endoscopic session will be performed at 3 months in both groups (repeat EB-RFA only in the EB-RFA arm). The primary endpoint is overall survival. Secondary endpoints include time to recurrent biliary obstruction, progression-free survival, adverse events, and technical/clinical success.

DETAILED DESCRIPTION:
Extrahepatic cholangiocarcinoma (eCCA) frequently presents as unresectable disease with obstructive jaundice. Although gemcitabine, cisplatin plus durvalumab (GCD) is the global standard first-line regimen, median overall survival remains approximately one year. Endobiliary radiofrequency ablation (EB-RFA) is biologically plausible to enhance local tumor control by inducing coagulative necrosis at the biliary stricture. Retrospective studies, including a multicenter dataset from participating institutions, suggest a survival benefit of repeated EB-RFA, especially when combined with systemic therapy. However, prospective randomized evidence is lacking.

This trial (BRAVE) randomizes eligible patients to EB-RFA plus standardized endoscopic stenting or endoscopic stenting alone, followed by GCD. A planned second endoscopic session is performed at Month 3 (window 2-4 months). Additional EB-RFA sessions (≥2-month intervals) are permitted in the EB-RFA arm if imaging shows potentially ablatable lesions and clinical benefit is expected.

The study aims to determine whether repeated EB-RFA prolongs survival and improves biliary patency when integrated with modern systemic therapy.

ELIGIBILITY:
Inclusion Criteria:

Histologically or cytologically confirmed extrahepatic cholangiocarcinoma (eCCA).

Unresectable disease (unresectable due to tumor/patient factors, or patient refusal of surgery).

Biliary obstruction requiring drainage, demonstrated by abnormal cholestatic liver tests, elevated bilirubin, radiologic evidence, or existing biliary drainage.

Planned initiation of first-line systemic therapy with durvalumab + gemcitabine + cisplatin (GCD).

Age ≥18 years.

Able to provide written informed consent.

Exclusion Criteria:

Prior radiotherapy or systemic therapy for the current eCCA.

Presence of a self-expanding metal stent that cannot be endoscopically removed.

Surgically altered anatomy except for Billroth-I; prior biliary reconstruction.

History of chronic cholangitis (e.g., primary sclerosing cholangitis, IgG4-related cholangitis).

Expected survival <3 months.

Inability to insert an oral endoscope or reach the papilla.

Contraindication to endobiliary RFA.

Pregnancy or possible pregnancy.

Any condition judged unsuitable by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-11-20 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | From randomization until death from any cause (up to 36 months after last enrollment)
  Overall survival is defined as the time from randomization to death from any cause. Participants still alive at the last confirmed contact will be censored at that date.

SECONDARY OUTCOMES:
Time to Recurrent Biliary Obstruction (TRBO) | From stent placement to RBO or censoring (up to 36 months)
  TRBO is defined as the time from stent placement to recurrent biliary obstruction (RBO).
Progression-Free Survival (PFS) | From randomization to radiologic progression or death (up to 36 months)
  Progression-free survival is defined per RECIST v1.1 based on imaging performed every 2-4 months.
Non-RBO Survival | Up to 36 months
  Time alive without recurrent biliary obstruction.
Survival Free From Late Biliary-Procedure-Related Adverse Events | Up to 36 months
  Late adverse events are defined as events occurring ≥15 days after the procedure (Tokyo Criteria 2024).
Incidence and Etiology of Recurrent Biliary Obstruction (RBO) | Up to 36 months
  Number and types of RBO events and their causes (sludge, tumor ingrowth/overgrowth, migration, dysfunction).
Early Adverse Events (≤14 days) | 14 days
  Procedure-related adverse events within 14 days, graded by Tokyo Criteria 2024.
Late Adverse Events (≥15 days) | Up to 36 months
  Procedure-related adverse events occurring ≥15 days post-procedure.
Technical Success | At index procedure
  Successful completion of the intended procedure:
  EB-RFA + plastic stent placement in the experimental arm
  Plastic stent placement in the comparator arm
Clinical Success | Within 14 days after stent placement
  Defined as:
  Hyperbilirubinemia: total bilirubin reduction ≥50% or ≤1.5 mg/dL within 14 days
  Others: normalization of ≥2 abnormal cholestatic/hepatocellular enzymes
  If baseline values are normal after prior drainage, absence of re-worsening beyond abnormal thresholds.
Number of RBO Events | Up to 36 months
  Count of recurrent biliary obstruction events per participant.
Number of Endoscopic Reinterventions | Up to 36 months
  Total number of endoscopic procedures including therapeutic interventions required during follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Tadahisa Inoue, Associate Professor, Principal Investigator — Department of Gastroenterology, Aichi Medical University; Jae Hee Cho, Professor, Principal Investigator — Department of Internal Medicine, Institute of Gastroenterology, Gangnam Severance Hospital, Yonsei University College of Medicine
Locations (8):
- Japan (4):
  - Aichi Medical University, Aichi
  - Nagoya City University Hospital, Aichi
  - Nagoya City University Midori Municipal Hospital, Aichi
  - Gifu University Hospital, Gifu
- South Korea (4):
  - Pusan National University Hospital, Busan
  - Gangnam Severance Hospital, Yonsei University College of Medicine, Seoul
  - Kangbuk Samsung Hospital, Sungkyunkwan University School of Medicine, Seoul
  - Severance Hospital, Yonsei University College of Medicine, Seoul

IPD SHARING:
Plan to Share IPD: No